CLINICAL TRIAL: NCT05245084
Title: An Open Label, Randomized, Single Dose, 2-sequence, 4-period, Cross-over Clinical Trial to Evaluate the Pharmacokinetics and Tolerability of CKD-386(3) With Co-administration of D013, D326, and D337 in Healthy Adult Volunteers
Brief Title: A Clinical Trial to Evaluate the Tolerability and Pharmacokinetics of CKD-386(3) 80/20/10mg
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A83_08BE2126
Record Dates: First submitted 2022-02-16; First posted 2022-02-17 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-01

CONDITIONS: Hypertension and Dyslipidemia
MeSH Terms: conditions — Hypertension; Dyslipidemias

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence 1 (Experimental): * Period 1: D013, D326, D337- A single oral dose of 3 tablets under fasting condition
  * Period 2: CKD-386(2)- A single oral dose of 1 tablet under fasting condition
  * Period 3: D013, D326, D337- A single oral dose of 3tablet s under fasting condition
  * Period 4: CKD-386(2)- A single oral dose of 1 tablet under fasting condition
  Interventions: Drug: CKD-386(3); Drug: D013, D326, D337
- Sequence 2 (Experimental): * Period 1: CKD-386(2)- A single oral dose of 1 tablet under fasting condition
  * Period 2: D013, D326, D337- A single oral dose of 3 tablets under fasting condition
  * Period 3: CKD-386(2)- A single oral dose of 1 tablet under fasting condition
  * Period 4: D013, D326, D337- A single oral dose of 3 tablets under fasting condition
  Interventions: Drug: CKD-386(3); Drug: D013, D326, D337

INTERVENTIONS:
Drug: CKD-386(3) — QD, PO
Drug: D013, D326, D337 — QD, PO

SUMMARY:
A Clinical Trial to evaluate the Pharmacokinetics and Tolerability of CKD-386(3)

DETAILED DESCRIPTION:
An open label, randomized, single dose, 2-sequence, 4-period, cross-over clinical trial to evaluate the pharmacokinetics and tolerability of CKD-386(3) with co-administration of D013, D326, and D337 in healthy adult volunteers

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult volunteers aged ≥ 19 years
2. Weight ≥50kg (man) or 45kg (woman), with calculated body mass index (BMI) of 18 to 30 kg/m2
3. Those who meet the blood pressure criteria during screening tests:

   * Systolic Blood Pressure: 90 to 139 mmHg
   * Diastolic Blood Pressure: 60 to 89 mmHg
4. Those who have no congenital diseases or chronic diseases and have no abnormal symptoms or findings.
5. Those who are eligible for clinical trials based on laboratory(hematology, blood chemistry, serology, urology) and 12-lead ECG results at screening.
6. Those who agree to contraception during the participation of clinical trial.
7. Individuals who voluntarily decide to participate and agree to comply with the cautions after fully understand the detailed description of this clinical trial.

Exclusion Criteria:

1. Those who received investigational products or participated in bioequivalence tests within 6 months before the first administration of clinical trial drugs.
2. Those who have used drugs that induce or inhibit drug metabolizing enzymes, such as barbiturates, within 1 month before the first dosing date, or who have used drugs that may interfere with this study within 10 days before the first dosing day (However, clinical investigational drugs) Participation is possible in consideration of pharmacokinetic and pharmacodynamic characteristics such as interaction with concomitant drugs and half-life of concomitant drugs)
3. Those who donated whole blood or apheresis within 8 weeks or 4 weeks respectfully, or received blood transfusion within a 4 weeks.
4. Those who have a history of gastrointestinal surgery except simple appendectomy and hernia surgery.
5. Those who exceed an alcohol and cigarette consumption than below criteria

   • Alcohol: Man_21 glasses/week, Woman_14 glasses/week (1 glass: Soju 50mL, Wine 30mL, or beer 250mL)

   • Heavy Smoking: 20 cigarettes/day
6. Patients with the following diseases

   * Patients with hypersensitivity to the main constituents or components of the investigational drug
   * Severe hepatic impairment, biliary atresia or cholestasis
   * Patients with hereditary angioedema or with a history of angioedema in the treatment of ACE inhibitors or angiotensin II receptor antagonists
   * Diabetes mellitus
   * Patients with moderate to severe renal impairment [glomerular filtration rate (eGFR) <60 mL / min / 1.73m^2]
   * Renal vascular hypertension patients
   * Patients with active liver disease, including unexplained persistent serum transaminase elevations or elevated serum transaminase elevations greater than three times the normal upper limit
   * Patients with myopathy or have a history of family or genetic history of myopathy
   * Hypothyroidism
   * If you have a history of muscle toxicity for other HMG-CoA converting enzymes or fibrate class drugs
7. Those who have genetic problems such as galactose intolerance, Lapp lactose deficiency or glucose-galactose malabsorption.
8. Those who are deemed insufficient to participate in this clinical study by investigators.
9. Woman who are pregnant or breastfeeding.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2022-06-06 (Actual); Study Completion 2022-06-20 (Actual)

PRIMARY OUTCOMES:
AUCt of CKD-386(3) | Pre-dose (0 hour), 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 8, 12, 24, 48, 72 hours
  Area under the concentration-time curve from time zero to time
Cmax of CKD-386(3) | Pre-dose (0 hour), 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 8, 12, 24, 48, 72 hours
  Maximum plasma concentration of the drug

CONTACTS AND LOCATIONS:
Overall Officials: Jaewoo Kim, M.D., Principal Investigator — Seoul, Gwanak-gu, South Korea, 08779
Locations (1):
- H plus Yangji hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No